CLINICAL TRIAL: NCT03077477
Title: Phase 1 Double-Blind, Placebo Controlled, Dose-Escalation Safety, Pharmacokinetic and Pharmacodynamic Study of Orally-Administered AMXT 1501 Dicaprate in Normal Healthy Volunteers
Brief Title: Study of Orally-Administered AMXT 1501 Dicaprate in Normal Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change in FDA required patient population decision prior to study start, new protocol developed, this protocol withdrawn
Sponsor: Aminex Therapeutics, Inc. (Industry)
Collaborators: Novella Clinical (Other); Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMXT1501-101
Record Dates: First submitted 2017-02-23; First posted 2017-03-13 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Neoplasms; Medication Toxicity; Tolerance
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: The study is comprised of a total of 8 cohorts; 4 single ascending dose (SAD) cohorts, 1 Food Effect (FE) Crossover cohort, and 3 multiple ascending dose (MAD) cohorts. Tablets will be administered after an overnight fast (10 hours) with at least 250 mL water. No food will be administered (exception for "fed" subjects, see below) for one hour thereafter.
  Each cohort will have a total 6 subjects: SAD and MAD (2 subjects receiving placebo and 4 subjects receiving active AMXT 1501 dicaprate); and FE crossover (6 subjects receiving active AMXT 1501 dicaprate).
Who Masked: Participant, Care Provider, Investigator
Masking Description: If subject is given active drug or placebo is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAD (Placebo Comparator): Cohort will have a total 6 subjects: SAD (2 subjects receiving placebo and 4 subjects receiving active AMXT 1501 dicaprate);
  SAD cohorts are defined as follows:
  * Cohort 1: One placebo and one AMXT 1501 dicaprate subject will be treated as sentinel subjects receiving one tablet each of their assigned treatment. Assuming no intolerance is noted after at least 3 days, the remaining cohort subjects (placebo, 1 subject and AMXT 1501 dicaprate, 3 subjects) will be treated.
  * Cohort 2: 2 subjects 2 placebo each and 4 subjects 2 AMXT 1501 dicaprate tablets each
  * Cohort 3: 2 subjects 4 placebos each and 4 subjects 4 AMXT 1501 dicaprate tablets each
  * Cohort 4: 2 subjects 8 placebos each and 4 subjects 8 AMXT 1501 dicaprate tablets each
  Interventions: Drug: AMXT 1501; Drug: Placebo Oral Tablet
- MAD (Placebo Comparator): Each cohort will have a total 6 subjects: MAD (2 subjects receiving placebo and 4 subjects receiving active AMXT 1501 dicaprate); MAD cohorts will receive dosing once daily for 14 consecutive days. Dosing will be contingent on adequate tolerance in Cohorts 1-5.
  * Cohort 6: 2 subjects 2 placebos each; 4 subjects 2 AMXT 1501 dicaprate tablets each
  * Cohort 7: 2 subjects 4 placebos each; 4 subjects 4 AMXT 1501 dicaprate tablets each
  * Cohort 8: 2 subjects 8 placebos each; 4 subjects 8 AMXT 1501 dicaprate tablets each
  Interventions: Drug: AMXT 1501; Drug: Placebo Oral Tablet
- FE (Active Comparator): Each cohort will have a total 6 subjects: FE crossover (6 subjects receiving active AMXT 1501 dicaprate).
  FE Crossover:
  • Cohort 5: 6 new subjects will be randomized to a fed (n=3 standard meal) or fasted (n=3) group and administered the highest dose of AMXT 1501 dicaprate tolerated by previous cohorts. First dose and accompanying assessments will be referred to as Period 1. Subjects will then crossover to the opposite diet plan (fed or fasted) and receive a second administration of study treatment at the same dose level. The second dose and assessments are referred to as Period 2. There will be a 7-day washout between doses administered in Periods 1 and 2.
  Interventions: Drug: AMXT 1501

INTERVENTIONS:
Drug: AMXT 1501 — Study treatment will be provided in tablet form; each containing 128 mg AMXT 1501 dicaprate salt, 80 mg of which is AMXT 1501 freebase (active drug), plus excipients and are orally administered.
  Other Names: AMX513
Drug: Placebo Oral Tablet — Reference Therapy, Dose and Route of Administration:
  Placebo Tablets, orally administered
  Arms: MAD; SAD

SUMMARY:
This is a Phase 1 study, which will assess the safety, PK, and pharmacodynamics (PD) of orally-administered AMXT 1501 dicaprate in normal healthy male volunteers.

The study is comprised of a total of 8 cohorts; 4 single ascending dose (SAD) cohorts, 1 Food Effect (FE) Crossover cohort, and 3 multiple ascending dose (MAD) cohorts. Tablets will be administered after an overnight fast (10 hours) with at least 250 mL water. No food will be administered (exception for "fed" subjects, see below) for one hour thereafter.

Each cohort will have a total 6 subjects: SAD and MAD (2 subjects receiving placebo and 4 subjects receiving active AMXT 1501 dicaprate); and FE crossover (6 subjects receiving active AMXT 1501 dicaprate).

DETAILED DESCRIPTION:
The Phase 1 study, which will assess the safety, PK, and pharmacodynamics (PD) of orally-administered AMXT 1501 dicaprate in normal healthy male volunteers.

The study is comprised of a total of 8 cohorts; 4 single ascending dose (SAD) cohorts, 1 Food Effect (FE) Crossover cohort, and 3 multiple ascending dose (MAD) cohorts. Tablets will be administered after an overnight fast (10 hours) with at least 250 mL water. No food will be administered (exception for "fed" subjects, see below) for one hour thereafter.

Each cohort will have a total 6 subjects: SAD and MAD (2 subjects receiving placebo and 4 subjects receiving active AMXT 1501 dicaprate); and FE crossover (6 subjects receiving active AMXT 1501 dicaprate).

SAD cohorts are defined as follows:

* Cohort 1: One placebo and one AMXT 1501 dicaprate subject will be treated as sentinel subjects receiving one tablet each of their assigned treatment. Assuming no intolerance is noted after at least 3 days, the remaining cohort subjects (placebo, 1 subject and AMXT 1501 dicaprate, 3 subjects) will be treated.
* Cohort 2: 2 subjects 2 placebo each and 4 subjects 2 AMXT 1501 dicaprate tablets each
* Cohort 3: 2 subjects 4 placebos each and 4 subjects 4 AMXT 1501 dicaprate tablets each
* Cohort 4: 2 subjects 8 placebos each and 4 subjects 8 AMXT 1501 dicaprate tablets each

FE Crossover:

• Cohort 5: 6 new subjects will be randomized to a fed (n=3 standard meal) or fasted (n=3) group and administered one dose lower of the maximum tolerated AMXT 1501 dose in the previous SAD cohorts. First dose and accompanying assessments will be referred to as Period 1. Subjects will then crossover to the opposite diet plan (fed or fasted) and receive a second administration of study treatment at the same dose level. The second dose and assessments are referred to as Period 2. There will be a 7-day washout between doses administered in Periods 1 and 2.

MAD cohorts will receive dosing once daily for 14 consecutive days. Dosing will be contingent on adequate tolerance in Cohorts 1-5.

* Cohort 6: 2 subjects 2 placebos each; 4 subjects 2 AMXT 1501 dicaprate tablets each
* Cohort 7: 2 subjects 4 placebos each; 4 subjects 4 AMXT 1501 dicaprate tablets each
* Cohort 8: 2 subjects 8 placebos each; 4 subjects 8 AMXT 1501 dicaprate tablets each

ELIGIBILITY:
Inclusion Criteria:

1. Adult males aged 18 to 55 years inclusive and between 18 to 30 kg/m2 body mass index (BMI).
2. Subjects who are healthy as determined by prestudy medical history, physical examination, and 12 Lead ECG.
3. Subjects whose clinical laboratory test results are not clinically relevant and are acceptable to the Investigator.
4. Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening.
5. Subjects who are negative for drugs of abuse and alcohol tests at screening and admission.
6. Subjects who are non-smokers for at least 1 month preceding screening.
7. Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

1. History of any important clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the study drug.
4. Subjects who have a history of relevant drug hypersensitivity to AMXT 1501.
5. Subjects who have a history of hearing loss.
6. Subjects who consume more than 21 units of alcohol a week. (unit = 1 glass of wine [125 mL] = 1 measure of spirits = ½ pint of beer)
7. Subjects who have a significant infection or known inflammatory process within 2 weeks of dosing or has febrile illness within 7 days of dosing.
8. Subjects who have acute gastrointestinal symptoms at the time of screening or admission (e.g. nausea, vomiting, diarrhea, heartburn).
9. Subjects who have an acute infection such as influenza at the time of screening or admission.
10. Subjects who do not agree to use medically acceptable methods of contraception during the study and for 90 days after the last dose of study drug
11. Subjects who use any medication including antacids, analgesics (with the exception of occasional use of up to 3 g of acetaminophen a day), herbal remedies (e.g., St. John's Wort), or vitamins and minerals from 2 weeks (for prescribed) or 1 week (for non-prescribed) prior to the first administration of study drug or longer if the medication has a long half-life. Occasional use of paracetamol/acetaminophen is allowed for minor pains and headache.
12. Subjects currently receiving medications or herbal supplements known to be potent inhibitors of CYP3A4 and potent inducers of CYP3A4 (from 2 weeks prior to the first administration of study drug). All subjects must avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer/inhibitory effects on CYP3A4.
13. Any intake of grapefruit, grapefruit juice, or other products containing grapefruit within 14 days of the first administration of study drug.
14. Subjects who have used any investigational drug in any clinical trial within 60 days of the screening visit.
15. Subjects who are vegans or have medical dietary restrictions.
16. Subjects who cannot communicate reliably with the Investigator.
17. Subjects who are unlikely to co-operate with the requirements of the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Determine the maximum feasible dose (MFD) | 6 months
  Determine the maximum feasible dose (MFD) of single and multiple doses of oral AMXT 1501 dicaprate in normal healthy volunteers.
Determine the pharmacokinetics (PK) of single and multiple by determining AUC | 6 months
  Determine the pharmacokinetics (PK) of single and multiple doses of oral AMXT 1501 dicaprate in normal subjects, by using Area under the plasma concentration versus time curve (AUC)
Determine the pharmacokinetics (PK) of single and multiple doses by determining Peak Plasma Concentration (Cmax) | 6 months
  Determine the pharmacokinetics (PK) of single and multiple doses of oral AMXT 1501 dicaprate in normal subjects, by using Peak Plasma Concentration (Cmax)
Assess influence of food on the PK by determining AUC | 6 months
  Assess influence of food on the PK of single doses of AMXT 1501 dicaprate, by comparing Area under the plasma concentration versus time curve (AUC)
Assess influence of food on the PK by determining Cmax | 6 months
  Assess influence of food on the PK of single doses of AMXT 1501 dicaprate, by comparing Peak Plasma Concentration (Cmax)

SECONDARY OUTCOMES:
To assess the effects of oral AMXT 1501 dicaprate on biomarkers to determine the appropriate dose level of the AMXT1501. | 8 months
  To assess the effects of oral AMXT 1501 by testing for the appropriate level of the drug measured by the biomarker Use the biomarker test level to determine the recommended AMXT1501 Phase 2 dose.

CONTACTS AND LOCATIONS:
Locations (1):
- IQVIA (formerly Quintiles IMS), Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD at this time